CLINICAL TRIAL: NCT04426695
Title: A Master Protocol Assessing the Safety, Tolerability, and Efficacy of Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies for the Treatment of Hospitalized Patients With COVID-19
Brief Title: Safety, Tolerability, and Efficacy of Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies for Hospitalized Adult Patients With COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2066; 2020-002537-15 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2); coronavirus; acute respiratory distress syndrome
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Distress Syndrome | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Intervention Model Description: Phase 1/Phase 2/Phase 3
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- On Low-Flow Oxygen (Experimental): Cohort 1 (C1): O2 saturation >93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device
  Interventions: Drug: REGN10933+REGN10987 combination therapy; Drug: Placebo
- With COVID-19 symptoms but not requiring supplemental O2 (Experimental): Cohort 1A (C1A): With COVID-19 symptoms but not requiring supplemental oxygen
  Interventions: Drug: REGN10933+REGN10987 combination therapy; Drug: Placebo
- High O2 No Mechanical Ventilation (Experimental): Cohort 2 (C2): On high-intensity oxygen (O2) therapy but not on mechanical ventilation
  Interventions: Drug: REGN10933+REGN10987 combination therapy; Drug: Placebo
- On Mechanical Ventilation (Experimental): Cohort 3 (C3): On mechanical ventilation
  Interventions: Drug: REGN10933+REGN10987 combination therapy; Drug: Placebo

INTERVENTIONS:
Drug: REGN10933+REGN10987 combination therapy — Administered intravenously (IV) single dose
  Other Names: REGN-COV2; REGEN-COV™; Ronapreve™; casirivimab; imdevimab
Drug: Placebo — Placebo IV Single Dose

SUMMARY:
The primary objectives are:

Pooled Phase 3 (Cohort 1) and Phase 2 (Cohort 1A)

* To evaluate the virologic efficacy of REGN10933+REGN10987 compared to placebo in reducing viral load of SARS-CoV-2
* To evaluate the clinical efficacy of REGN10933+REGN10987 compared to placebo, as measured by death or mechanical ventilation

Phase 1/2 (Cohort 1)

* To exclude futility of REGN10933+REGN10987 compared to placebo, as measured by death or mechanical ventilation
* To evaluate the safety and tolerability of REGN10933+REGN10987 compared to placebo

ELIGIBILITY:
Key Inclusion Criteria:

* Has SARS-CoV-2-positive antigen or molecular diagnostic test (by validated SARS-CoV-2 antigen, RT-PCR, or other molecular diagnostic assay, using an appropriate sample such as NP, nasal, oropharyngeal [OP], or saliva) ≤72 hours prior to randomization and no alternative explanation for current clinical condition. A historical record of positive result from test conducted ≤72 hours prior to randomization is acceptable.
* Has symptoms consistent with COVID-19, as determined by investigator, with onset ≤10 days before randomization
* Hospitalized for ≤72 hours with at least 1 of the following at randomization; patients meeting more than one criterion will be categorized in the most severely affected category:

  1. Cohort 1A: With COVID-19 symptoms but not requiring supplemental oxygen
  2. Cohort 1: Maintains O2 saturation >93% on low-flow oxygen as defined in the protocol
  3. Cohort 2: High-intensity oxygen therapy without mechanical ventilation as defined in the protocol
  4. Cohort 3: On mechanical ventilation

Key Exclusion Criteria:

* Phase 1 Only: Patients maintaining O2 saturation >94% on room air
* In the opinion of the investigator, unlikely to survive for >48 hours from screening
* Receiving extracorporeal membrane oxygenation (ECMO)
* Has new-onset stroke or seizure disorder during hospitalization
* Initiated on renal replacement therapy due to COVID-19

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2252 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (101):
- United States (76):
  - Regeneron Study Site, Birmingham, Alabama
  - Regeneron Study Site, Chandler, Arizona
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site 1, Tucson, Arizona
  - Regeneron Study Site, Long Beach, California
  - Regeneron Study Site, Mission Hills, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, Santa Monica, California
  - Regeneron Study Site, Stanford, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, Boca Raton, Florida
  - Regeneron Study Site, Ft. Pierce, Florida
  - Regeneron Study Site, Gainesville, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Pensacola, Florida
  - Regeneron Study Site, Sarasota, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Augusta, Georgia
  - Regeneron Study Site, Marietta, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Glenview, Illinois
  - Regeneron Study Site, Urbana, Illinois
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Louisville, Kentucky
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Grand Rapids, Michigan
  - Regeneron Study Site, Royal Oak, Michigan
  - Regeneron Study Site, Rochester, Minnesota
  - Regeneron Study Site, Chesterfield, Missouri
  - Regeneron Study Site, St Louis, Missouri
  - Regeneron Study Site, Omaha, Nebraska
  - Regeneron Study Site, Las Vegas, Nevada
  - Regeneron Study Site, Englewood, New Jersey
  - Regeneron Study Site, Hackensack, New Jersey
  - Regeneron Study Site, Morristown, New Jersey
  - Regeneron Study Site, Neptune City, New Jersey
  - Regeneron Study Site, Pennington, New Jersey
  - Regeneron Study Site, Summit, New Jersey
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, Albuquerque, New Mexico
  - Regeneron Study Site, Brooklyn, New York
  - Regeneron Study Site, Buffalo, New York
  - Regeneron Study Site 1, Buffalo, New York
  - Regeneron Study Site 2, Buffalo, New York
  - Regeneron Study Site, Jamaica, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Rochester, New York
  - Regeneron Study Site, Syracuse, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, West Islip, New York
  - Regeneron Study Site, White Plains, New York
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, Greensboro, North Carolina
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Providence, Rhode Island
  - Regeneron Study Site, Sioux Falls, South Dakota
  - Regeneron Study Site 1, Amarillo, Texas
  - Regeneron Study Site 2, Amarillo, Texas
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Lubbock, Texas
  - Regeneron Study Site, Sugar Land, Texas
  - Regeneron Study Site, Tyler, Texas
  - Regeneron Study Site, Murray, Utah
  - Regeneron Study Site, Salt Lake City, Utah
  - Regeneron Study Site, Richmond, Virginia
  - Regeneron Study Site, Everett, Washington
  - Regeneron Study Site 1, Seattle, Washington
  - Regeneron Study Site, Madison, Wisconsin
- Brazil (10):
  - Regeneron Study Site, Fortaleza, Ceará
  - Regeneron Study Site, Salvador, Estado de Bahia
  - Regeneron Study Site, Curitiba, Paraná
  - Regeneron Study Site, Passo Fundo, Rio Grande do Sul
  - Regeneron Study Site, Porto Alegre, Rio Grande do Sul
  - Regeneron Study Site, Chapecó, Santa Catarina
  - Regeneron Study Site, Criciúma, Santa Catarina
  - Regeneron Study Site, Botucatu, São Paulo
  - Regeneron Study Site, Campinas, São Paulo
  - Regeneron Study Site, São Paulo
- Chile (4):
  - Regeneron Study Site 1, Las Condes, Santiago de Chile
  - Regeneron Study Site 2, Las Condes, Santiago de Chile
  - Regeneron Study Site, Vitacura, Santiago de Chile
  - Regeneron Study Site, Santiago
- Mexico (9):
  - Regeneron Study Site, Guadalajara, Jalisco
  - Regeneron Study Site, Monterrey, Nuevo León
  - Regeneron Study Site, Culiacán, Sinaloa
  - Regeneron Study Site, Culiacán
  - Regeneron Study Site 1, Mérida
  - Regeneron Study Site 2, Mérida
  - Regeneron Study Site, Monterrey
  - Regeneron Study Site, Veracruz
  - Regeneron Study Site, Zapopan
- Regeneron Study Site, Chisinau, Moldova
- Regeneron Study Site, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., Food and Drug Administration (FDA), European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Somersan-Karakaya S, Mylonakis E, Mou J, Oviedo-Orta E, O'Brien MP, Mas Casullo V, Mahmood A, Hooper AT, Hussein M, Ali S, Marty FM, Forleo-Neto E, Bhore R, Hamilton JD, Herman GA, Hirshberg B, Weinreich DM. Effectiveness of Casirivimab and Imdevimab Antibody Combination in Immunocompromised Hospitalized Patients With Coronavirus Disease 2019: A Post Hoc Analysis in a Phase 1/2/3 Double-Blind Trial. Open Forum Infect Dis. 2023 Apr 19;10(5):ofad211. doi: 10.1093/ofid/ofad211. eCollection 2023 May. PMID 37229174
- [Derived] Hooper AT, Somersan-Karakaya S, McCarthy SE, Mylonakis E, Ali S, Mei J, Bhore R, Mahmood A, Geba GP, Dakin P, Weinreich DM, Yancopoulos GD, Herman GA, Hamilton JD; COVID-19 Phase 2/3 Hospitalized Trial Team. Casirivimab and Imdevimab Treatment Reduces Viral Load and Improves Clinical Outcomes in Seropositive Hospitalized COVID-19 Patients with Nonneutralizing or Borderline Neutralizing Antibodies. mBio. 2022 Dec 20;13(6):e0169922. doi: 10.1128/mbio.01699-22. Epub 2022 Oct 18. PMID 36255239
- [Derived] Somersan-Karakaya S, Mylonakis E, Menon VP, Wells JC, Ali S, Sivapalasingam S, Sun Y, Bhore R, Mei J, Miller J, Cupelli L, Forleo-Neto E, Hooper AT, Hamilton JD, Pan C, Pham V, Zhao Y, Hosain R, Mahmood A, Davis JD, Turner KC, Kim Y, Cook A, Kowal B, Soo Y, DiCioccio AT, Geba GP, Stahl N, Lipsich L, Braunstein N, Herman GA, Yancopoulos GD, Weinreich DM; COVID-19 Phase 2/3 Hospitalized Trial Team. Casirivimab and Imdevimab for the Treatment of Hospitalized Patients With COVID-19. J Infect Dis. 2022 Dec 28;227(1):23-34. doi: 10.1093/infdis/jiac320. PMID 35895508
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2324 participants were screened and 2203 participants randomized and treated, 49 participants were randomized but not treated, and 72 discontinued at the screening phase. Reasons for discontinuation at screening phase: 54 - Screen Failure, 10 - Subject Decision, 1- Sponsor Request, 7- Other.
Groups:
- Phase 1: Cohort 1 (Placebo): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 1: Cohort 1 (R10933+R10987 2400 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 milligrams (mg) intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 1: Cohort 1 (R10933+R10987 8000 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 2: Cohort 1 (Placebo): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 1)
- Phase 2: Cohort 1 (R10933+R10987 2400 mg: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 milligrams (mg) intravenously on Day 1 in Phase 2 (Cohort 1)
- Phase 2: Cohort 1 (R10933+R10987 8000 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 1)
- Phase 3: Cohort 1 (Placebo): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 3 (Cohort 1)
- Phase 3: Cohort 1 (R10933+R10987 2400 mg): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 milligrams (mg) intravenously on Day 1 in Phase 3 (Cohort 1)
- Phase 3: Cohort 1 (R10933+R10987 8000 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 3 (Cohort 1)
- Phase 2: Cohort 1A (Placebo): Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2: Cohort 1A (R10933+R10987 2400 mg IV): Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2: Cohort 1A (R10933+R10987 8000 mg IV): Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2: Cohort 2 (Placebo): Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2: Cohort 2 (R10933+R10987 2400 mg IV): Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2: Cohort 2 (R10933+R10987 8000 mg IV): Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2: Cohort 3 (Placebo): Participants on mechanical ventilation received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 2: Cohort 3 (R10933+R10987 2400 mg IV): Participants on mechanical ventilation received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 2: Cohort 3 (R10933+R10987 8000 mg IV): Participants on mechanical ventilation received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 3).
Period: Overall Study
Arm/Group | Phase 1: Cohort 1 (Placebo) | Phase 1: Cohort 1 (R10933+R10987 2400 mg IV) | Phase 1: Cohort 1 (R10933+R10987 8000 mg IV) | Phase 2: Cohort 1 (Placebo) | Phase 2: Cohort 1 (R10933+R10987 2400 mg | Phase 2: Cohort 1 (R10933+R10987 8000 mg IV) | Phase 3: Cohort 1 (Placebo) | Phase 3: Cohort 1 (R10933+R10987 2400 mg) | Phase 3: Cohort 1 (R10933+R10987 8000 mg IV) | Phase 2: Cohort 1A (Placebo) | Phase 2: Cohort 1A (R10933+R10987 2400 mg IV) | Phase 2: Cohort 1A (R10933+R10987 8000 mg IV) | Phase 2: Cohort 2 (Placebo) | Phase 2: Cohort 2 (R10933+R10987 2400 mg IV) | Phase 2: Cohort 2 (R10933+R10987 8000 mg IV) | Phase 2: Cohort 3 (Placebo) | Phase 2: Cohort 3 (R10933+R10987 2400 mg IV) | Phase 2: Cohort 3 (R10933+R10987 8000 mg IV)
Started | 21 | 19 | 20 | 208 | 211 | 210 | 251 | 252 | 252 | 201 | 205 | 203 | 52 | 58 | 54 | 12 | 12 | 11
Treated | 18 | 18 | 20 | 204 | 206 | 205 | 247 | 246 | 246 | 198 | 202 | 197 | 51 | 56 | 54 | 12 | 12 | 11
Completed | 13 | 12 | 16 | 146 | 153 | 148 | 186 | 195 | 189 | 157 | 165 | 166 | 33 | 28 | 31 | 5 | 4 | 7
Not Completed | 8 | 7 | 4 | 62 | 58 | 62 | 65 | 57 | 63 | 44 | 40 | 37 | 19 | 30 | 23 | 7 | 8 | 4
Not completed — Death | 2 | 0 | 1 | 27 | 25 | 21 | 42 | 23 | 37 | 14 | 8 | 7 | 13 | 25 | 19 | 7 | 8 | 4
Not completed — Lost to Follow-up | 2 | 4 | 1 | 19 | 10 | 14 | 5 | 14 | 10 | 11 | 12 | 6 | 2 | 2 | 2 | 0 | 0 | 0
Not completed — Participant Decision | 1 | 2 | 2 | 12 | 18 | 22 | 13 | 13 | 10 | 15 | 16 | 17 | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Request | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but Never Treated | 3 | 1 | 0 | 4 | 5 | 5 | 4 | 6 | 6 | 3 | 3 | 6 | 1 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least one dose (full or partial) of the study drug.
Groups:
- Phase 1: Cohort 1 (R10933+R10987 2400 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 1 (Cohort 1)
- Phase 2: Cohort 1 (R10933+R10987 2400 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 1)
- Phase 3: Cohort 1 (R10933+R10987 2400 mg IV): Phase 1: Cohort 1 (R10933+R10987 2400 mg IV)Edit Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cohort 1 (Placebo) | Phase 1: Cohort 1 (R10933+R10987 2400 mg IV) | Phase 1: Cohort 1 (R10933+R10987 8000 mg IV) | Phase 2: Cohort 1 (Placebo) | Phase 2: Cohort 1 (R10933+R10987 2400 mg IV) | Phase 2: Cohort 1 (R10933+R10987 8000 mg IV) | Phase 3: Cohort 1 (Placebo) | Phase 3: Cohort 1 (R10933+R10987 2400 mg IV) | Phase 3: Cohort 1 (R10933+R10987 8000 mg IV) | Phase 2: Cohort 1A (Placebo) | Phase 2: Cohort 1A (R10933+R10987 2400 mg IV) | Phase 2: Cohort 1A (R10933+R10987 8000 mg IV) | Phase 2: Cohort 2 (Placebo) | Phase 2: Cohort 2 (R10933+R10987 2400 mg IV) | Phase 2: Cohort 2 (R10933+R10987 8000 mg IV) | Phase 2: Cohort 3 (Placebo) | Phase 2: Cohort 3 (R10933+R10987 2400 mg IV) | Phase 2: Cohort 3 (R10933+R10987 8000 mg IV) | Total
Number analyzed (Participants) | 18 | 18 | 20 | 204 | 206 | 205 | 247 | 246 | 246 | 198 | 202 | 197 | 51 | 56 | 54 | 12 | 12 | 11 | 2203
Age, Customized [Count of Participants; unit: Participants]
  Age: 18- <40 years | 1 | 1 | 2 | 26 | 16 | 17 | 29 | 28 | 14 | 22 | 20 | 20 | 4 | 4 | 6 | 0 | 1 | 1 | 212
  Age: 40- <65 years | 9 | 8 | 10 | 82 | 99 | 96 | 105 | 119 | 127 | 82 | 101 | 91 | 30 | 23 | 24 | 6 | 4 | 5 | 1021
  Age: >=65 years | 8 | 9 | 8 | 96 | 91 | 92 | 113 | 99 | 105 | 94 | 81 | 86 | 17 | 29 | 24 | 6 | 7 | 5 | 970
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 10 | 90 | 98 | 98 | 113 | 112 | 115 | 91 | 87 | 89 | 17 | 20 | 20 | 8 | 4 | 2 | 990
  Male | 10 | 10 | 10 | 114 | 108 | 107 | 134 | 134 | 131 | 107 | 115 | 108 | 34 | 36 | 34 | 4 | 8 | 9 | 1213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 10 | 49 | 50 | 52 | 92 | 94 | 82 | 38 | 53 | 40 | 13 | 22 | 18 | 6 | 5 | 4 | 647
  Not Hispanic or Latino | 6 | 11 | 10 | 144 | 148 | 146 | 146 | 140 | 155 | 148 | 138 | 143 | 35 | 33 | 30 | 6 | 7 | 7 | 1453
  Unknown or Not Reported | 0 | 0 | 0 | 11 | 8 | 7 | 9 | 12 | 9 | 12 | 11 | 14 | 3 | 1 | 6 | 0 | 0 | 0 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 2 | 9 | 9 | 13 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 36
  Asian | 0 | 2 | 0 | 6 | 7 | 6 | 6 | 10 | 9 | 11 | 8 | 6 | 2 | 2 | 1 | 1 | 1 | 0 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 10
  Black or African American | 3 | 2 | 8 | 34 | 21 | 33 | 26 | 32 | 25 | 27 | 32 | 25 | 7 | 6 | 9 | 1 | 1 | 3 | 295
  White | 12 | 11 | 11 | 136 | 146 | 134 | 159 | 151 | 158 | 111 | 116 | 131 | 33 | 39 | 36 | 8 | 9 | 5 | 1406
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 1 | 25 | 30 | 29 | 47 | 43 | 40 | 49 | 46 | 34 | 7 | 8 | 8 | 1 | 1 | 3 | 378

OUTCOME MEASURES:

1. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Time-weighted Average (TWA) Change in Viral Load in Nasopharyngeal (NP) Samples Based on Seronegative mFAS
Description: Time-weighted average daily change from Day 1 to Day 7 in viral load (log10 copies/mL), as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Day 1 to Day 7
Population: The seronegative modified full analysis set (mFAS) was defined as all participants in mFAS with documented seronegative status at the baseline. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Least Squares Mean (Standard Error); unit: log10 copies/milliliter (mL)
Groups:
- Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 3 (Cohort 1) and participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of matching placebo intravenously on Day 1 in Phase 2 (Cohort 1A).
- Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (2400 mg) intravenously on Day 1 in Phase 3 (Cohort 1) and participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 (2400 mg) intravenously on Day 1 in Phase 2 (Cohort 1A).
- Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (8000 mg) intravenously on Day 1 in Phase 3 (Cohort 1) and participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 (8000 mg) intravenously on Day 1 in Phase 2 (Cohort 1A).
- Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (2400 mg and 8000 mg) intravenously on Day 1 in Phase 3 (Cohort 1) and participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 (2400 mg and 8000 mg) intravenously on Day 1 in Phase 2 (Cohort 1A).
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 131 | 150 | 160 | 310
log10 copies/milliliter (mL) | -1.03 (0.10) | -1.28 (0.09) | -1.34 (0.09) | -1.31 (0.06)
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0663, ANCOVA — P-value for change from baseline on log scale for each treatment group was based on the Analysis of covariance (ANCOVA) model with treatment group; Least Square (LS) Mean Difference = -0.25, 95% CI 2-sided [-0.51 to 0.02]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0204, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = -0.31, 95% CI [-0.57 to 0.05]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; To control alpha at a strict 0.05 level, this endpoint was tested hierarchically, with the virologic endpoint tested first. All hierarchical testing was done using the combined dose group; Test type: Superiority; p = 0.0172, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = -0.28, 95% CI 2-sided [-0.51 to -0.05]

2. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Percentage of Participants Who Died or Went on Mechanical Ventilation From Day 6 Through Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who died or went on mechanical ventilation from Day 6 through Day 29 based on high viral load mFAS were reported.
Time Frame: Day 6 to Day 29
Population: The High Viral Load mFAS was defined as all participants in mFAS with baseline SARS-CoV-2 viral load greater than (>) 10^6 copies per milliliter (mL). Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 211 | 220 | 225 | 445
Percentage of Participants | 13.3 [9.0 to 18.6] | 7.3 [4.2 to 11.5] | 12.4 [8.4 to 17.5] | 9.9 [7.3 to 13.0]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0431, Cochran-Mantel-Haenszel — P-value was derived Cochran-Mantel-Haenszel (CMH) test stratified by the type of background standard-of-care (antiviral therapies and non-antiviral therapies). If np < =5 or n(1-p) <= 5 in any treatment group, p-value was based on Fisher Exact Test
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.7975, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.2048, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

3. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Percentage of Participants Who Died or Went on Mechanical Ventilation From Day 6 Through Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died or went on mechanical ventilation from Day 6 through Day 29 based on seronegative mFAS were reported.
Time Frame: Day 6 to Day 29
Population: The seronegative mFAS was defined as all participants in mFAS with documented seronegative status at the baseline. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 147 | 162 | 179 | 341
Percentage of Participants | 15.0 [9.6 to 21.8] | 4.9 [2.2 to 9.5] | 10.6 [6.5 to 16.1] | 7.9 [5.3 to 11.3]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0039, Cochran-Mantel-Haenszel — P-value was derived CMH test stratified by the type of background standard-of-care (antiviral therapies and non-antiviral therapies). If np < =5 or n(1-p) <= 5 in any treatment group, p-value was based on Fisher Exact Test
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.2415, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0195, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

4. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Percentage of Participants Who Died or Went on Mechanical Ventilation From Day 6 Through Day 29 Based on Overall mFAS
Description: Percentage of participants who died or went on mechanical ventilation from Day 6 through Day 29 based on overall FAS were reported.
Time Frame: Day 6 to Day 29
Population: The mFAS included all FAS participants with a positive SARS-CoV-2 RT-qPCR conducted in the central laboratory in NP swab samples at randomization. Analysis based on treatment allocated (as randomized). "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 367 | 387 | 383 | 770
Percentage of Participants | 10.6 [7.7 to 14.2] | 5.4 [3.4 to 8.2] | 10.7 [7.8 to 14.2] | 8.1 [6.2 to 10.2]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0085, Cochran-Mantel-Haenszel — P-value was derived CMH test stratified by the type of background standard-of-care (antiviral therapies and non-antiviral therapies). If np < = 5 or n(1-p) <= 5 in any treatment group, p-value is based on Fisher Exact Test
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.9902, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.1486, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]

5. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Percentage of Participants Who Died or Went on Mechanical Ventilation From Day 1 Through Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who died or went on mechanical ventilation from Day 1 through Day 29 based on high viral load mFAS were reported.
Time Frame: Day 1 to Day 29
Population: The High Viral Load mFAS was defined as all participants in mFAS with baseline SARS-CoV-2 viral load > 10^6 copies per mL. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 229 | 231 | 236 | 467
Percentage of Participants | 18.8 [13.9 to 24.4] | 10.0 [6.4 to 14.6] | 14.4 [10.2 to 19.5] | 12.2 [9.4 to 15.5]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0092, Cochran-Mantel-Haenszel — P-value was derived CMH test stratified by the type of background standard-of-care (antiviral therapies and non-antiviral therapies). If np < = 5 or n(1-p) <= 5 in any treatment group, p-value was based on Fisher Exact Test
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.2210, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0249, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]

6. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Percentage of Participants Who Died or Went on Mechanical Ventilation From Day 1 Through Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died or went on mechanical ventilation from Day 1 through Day 29 based on seronegative mFAS were reported.
Time Frame: Day 1 to Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 160 | 172 | 188 | 360
Percentage of Participants | 19.4 [13.6 to 26.4] | 8.1 [4.5 to 13.3] | 12.2 [7.9 to 17.8] | 10.3 [7.3 to 13.9]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0045, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0714, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0061, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]

7. Primary Outcome: Pooled Analysis (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Percentage of Participants Who Died or Went on Mechanical Ventilation From Day 1 Through Day 29 Based on Overall mFAS
Description: Percentage of participants who died or went on mechanical ventilation from Day 1 through Day 29 based on overall mFAS were reported.
Time Frame: Day 1 to Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 393 | 406 | 398 | 804
Percentage of Participants | 14.8 [11.4 to 18.7] | 7.9 [5.5 to 10.9] | 12.6 [9.5 to 16.2] | 10.2 [8.2 to 12.5]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0023, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.3544, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0212, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]

8. Primary Outcome: Pooled Analysis (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Number of Participants With Treatment-Emergent Serious Adverse Events
Description: Treatment-emergent adverse events are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the observation period.
Time Frame: Up to Day 169
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching R10933+R10987 intravenously on Day 1
- Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (2400 mg) intravenously on Day 1
- Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (8000 mg) intravenously on Day 1
- Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (2400 mg and 8000 mg) intravenously on Day 1
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 222 | 224 | 225 | 449
Participants | 54 | 45 | 47 | 92

9. Primary Outcome: Pooled Analysis (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Number of Participants With Grade >=2 Infusion Related Reactions up to Day 4
Description: Infusion-related reactions are defined as any relevant adverse event that occurs during the infusion or up to day 4. The severity of adverse events (including test findings classified as adverse events) were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).
Time Frame: Up to Day 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 222 | 224 | 225 | 449
Participants | 3 | 2 | 6 | 8

10. Primary Outcome: Pooled Analysis (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Number of Participants With Grade >=2 Hypersensitivity Reactions Up to Day 29
Description: Hypersensitivity reactions are defined as any relevant adverse event that occurs during the infusion or up to study day 29. The severity of adverse events (including test findings classified as adverse events) were graded according to NCI-CTCAE.
Time Frame: Up to Day 29
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 222 | 224 | 225 | 449
Participants | 1 | 2 | 2 | 4

11. Primary Outcome: Pooled Analysis (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Cumulative Incidence of Death or Mechanical Ventilation Based on Seronegative mFAS
Description: Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: Up to Day 29
Population: Seronegative modified full analysis set (mFAS) was defined as all participants in mFAS with documented seronegative status at the baseline. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 1 [Cohort 1] and Phase 2 [Cohort 1].
Measure: Number (80% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 32 | 46 | 41 | 87
Cumulative Incidence Percentage | 23.0 [16.9 to 30.9] | 15.1 [10.5 to 21.4] | 20.3 [14.7 to 27.8] | 17.6 [13.8 to 22.3]

12. Primary Outcome: Pooled Analysis (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Cumulative Incidence of Death or Mechanical Ventilation Based on High Viral Load mFAS
Description: Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: Up to Day 29
Population: High Viral Load mFAS was defined as all participants in mFAS with baseline SARS-CoV-2 viral load greater than (>) 10^6 copies per milliliter (mL). As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 1 [Cohort 1] and Phase 2 [Cohort 1].
Measure: Number (80% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 50 | 53 | 58 | 111
Cumulative Incidence Percentage | 20.7 [15.7 to 26.9] | 18.9 [14.3 to 24.8] | 11.6 [8.0 to 16.8] | 15.3 [12.2 to 19.0]

13. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Went on Mechanical Ventilation by Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who went on mechanical ventilation by Day 29 based on High Viral Load mFAS in pooled analysis phase 3 (Cohort 1) and phase 2 (Cohort 1A) was reported.
Time Frame: by Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 229 | 231 | 236 | 467
Percentage of Participants | 11.4 [7.6 to 16.2] | 6.1 [3.4 to 10.0] | 8.5 [5.3 to 12.8] | 7.3 [5.1 to 10.0]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0575, Cochran-Mantel-Haenszel — P-value is derived Cochran-Mantel-Haenszel (CMH) test stratified by the type of background standard-of-care (antiviral therapies and non-antiviral therapies). If np < =5 or n(1-p) <= 5 in any treatment group, p-value is based on Fisher Exact Test
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.3133, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0849, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

14. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Went on Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Description: Percentage of participants who went on mechanical ventilation at Day 29 based on Seronegative mFAS in pooled analysis phase 3 (Cohort 1) and phase 2 (Cohort 1A) was reported.
Time Frame: by Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 160 | 172 | 188 | 360
Percentage of Participants | 10.0 [5.8 to 15.7] | 5.8 [2.8 to 10.4] | 7.4 [4.1 to 12.2] | 6.7 [4.3 to 9.8]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.2167, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.4123, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.2206, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

15. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 6 Through Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who died from Day 6 through Day 29 based on high viral load mFAS were reported.
Time Frame: Day 6 to Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 222 | 226 | 228 | 454
Percentage of Participants | 13.1 [8.9 to 18.2] | 7.1 [4.1 to 11.2] | 10.1 [6.5 to 14.8] | 8.6 [6.2 to 11.6]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0383, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.3296, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0766, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

16. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 6 Through Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died from Day 6 through Day 29 Based on seronegative mFAS in pooled analysis phase 3 (cohort 1) and phase 2 (cohort 1A) were reported.
Time Frame: Day 6 to Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 153 | 167 | 181 | 348
Percentage of Participants | 13.7 [8.7 to 20.2] | 4.8 [2.1 to 9.2] | 7.2 [3.9 to 12.0] | 6.0 [3.8 to 9.1]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0070, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0507, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0051, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

17. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 1 Through Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who died from Day 1 through Day 29 based on High Viral Load mFAS in pooled analysis phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported.
Time Frame: Day 1 to Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 229 | 231 | 236 | 467
Percentage of participants | 14.4 [10.1 to 19.6] | 7.4 [4.3 to 11.5] | 11.0 [7.3 to 15.7] | 9.2 [6.7 to 12.2]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0174, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.2900, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0454, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

18. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 1 Through Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died from Day 1 through Day 29 based on seronegative mFAS in pooled analysis phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported.
Time Frame: Day 1 to Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 160 | 172 | 188 | 360
Percentage of Participants | 15.0 [9.9 to 21.5] | 5.2 [2.4 to 9.7] | 8.0 [4.5 to 12.8] | 6.7 [4.3 to 9.8]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0040, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0413, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0032, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

19. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Were Discharged by Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who were discharged by Day 29 based on High Viral Load mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) were reported.
Time Frame: by Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 229 | 231 | 236 | 467
Percentage of Participants | 80.3 [74.6 to 85.3] | 89.2 [84.4 to 92.9] | 86.9 [81.9 to 90.9] | 88.0 [84.7 to 90.8]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0105, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0622, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0088, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

20. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Were Discharged by Day 29 Based on Seronegative mFAS
Description: Percentage of participants who were discharged by Day 29 based on seronegative mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) were reported.
Time Frame: by Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 160 | 172 | 188 | 360
Percentage of Participants | 81.3 [74.3 to 87.0] | 90.1 [84.6 to 94.1] | 89.9 [84.7 to 93.8] | 90.0 [86.4 to 92.9]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0275, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0223, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0072, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

21. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died or Were Readmitted to Hospital Over Time Based on High Viral Load mFAS
Description: Percentage of participants who died or were readmitted to hospital over time based on High Viral Load mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A)were reported. Readmission to hospital was based on investigator report.
Time Frame: Up to Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 229 | 231 | 236 | 467
Percentage of Participants | 21.0 [15.9 to 26.8] | 15.2 [10.8 to 20.4] | 17.4 [12.8 to 22.8] | 16.3 [13.0 to 19.9]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.1032, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.3350, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.1314, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

22. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died or Were Readmitted to Hospital by Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died or were readmitted to hospital at Day 29 based on seronegative mFAS in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported. Readmission to hospital was based on investigator report.
Time Frame: by Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 160 | 172 | 188 | 360
Percentage of Participants | 24.4 [17.9 to 31.8] | 11.6 [7.2 to 17.4] | 12.8 [8.4 to 18.4] | 12.2 [9.0 to 16.1]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.00024, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0054, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

23. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death (ie, Overall Survival) by Day 29 Based on High Viral Load mFAS
Description: Overall Survival was defined as time interval from randomization to death. Percentage of participants with cumulative incidence of death (ie, overall survival) at Day 29 from randomization based on High Viral Load mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 181 | 201 | 190 | 391
Cumulative Incidence Percentage | 14.9 [10.8 to 20.3] | 7.7 [4.8 to 12.1] | 11.7 [8.1 to 16.7] | 9.7 [7.3 to 12.9]

24. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death (ie, Overall Survival) by Day 29 Based on Seronegative mFAS
Description: Overall Survival was defined as time interval from randomization to death. Percentage of participants with cumulative incidence of death (ie, overall survival) at Day 29 from randomization based on seronegative mFAS in phase 3 (Cohort 1) and phase 2 (Cohort 1A)were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 121 | 148 | 160 | 308
Cumulative Incidence Percentage | 15.8 [10.9 to 22.7] | 5.6 [3.0 to 10.5] | 8.4 [5.1 to 13.5] | 7.0 [4.8 to 10.3]

25. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Mechanical Ventilation by Day 29 Based on High Viral Load mFAS
Description: Number of participants with cumulative incidence of mechanical ventilation by Day 29 based on High Viral Load mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 170 | 194 | 183 | 377
Cumulative Incidence Percentage | 11.8 [8.2 to 16.8] | 6.3 [3.7 to 10.3] | 9.1 [6.0 to 13.8] | 7.7 [5.5 to 10.6]

26. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Description: Percentage of participants with cumulative incidence of mechanical ventilation by Day 29 based on seronegative mFAS in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 114 | 143 | 152 | 295
Cumulative Incidence Percentage | 10.6 [6.6 to 16.8] | 6.0 [3.3 to 11.0] | 7.9 [4.8 to 13.0] | 7.0 [4.8 to 10.3]

27. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death or Mechanical Ventilation by Day 29 Based on High Viral Load mFAS
Description: Percentage of participants with cumulative incidence of death or mechanical ventilation by Day 29 based on High Viral Load mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 170 | 194 | 183 | 377
Cumulative Incidence Percentage | 19.1 [14.6 to 24.9] | 10.2 [6.9 to 15.0] | 15.0 [11.0 to 20.4] | 12.7 [9.9 to 16.1]

28. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death or Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Description: Percentage of participants with cumulative incidence of death or mechanical ventilation by Day 29 based on seronegative mFAS in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 114 | 143 | 152 | 295
Cumulative Incidence Percentage | 20.1 [14.6 to 27.3] | 8.4 [5.1 to 13.8] | 12.7 [8.7 to 18.6] | 10.7 [7.9 to 14.5]

29. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Time to Discharge From Hospital Based on High Viral Load mFAS
Description: Time to discharge from hospital based on High Viral Load mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) was reported.
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 229 | 231 | 236 | 467
Days | 5.0 [4.0 to 6.0] | 4.0 [4.0 to 5.0] | 4.0 [3.0 to 5.0] | 4.0 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0533, Log Rank — P-value based on stratified log-rank test with the type of background standard-of-care and baseline serostatus as stratification factors
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0411, Log Rank — [p-value comment as in outcome 29, analysis 1]
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0229, Log Rank — [p-value comment as in outcome 29, analysis 1]

30. Secondary Outcome: Pooled Analysis Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Time to Discharge From Hospital Based on Seronegative mFAS
Description: Time to discharge from hospital based on Seronegative mFAS in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) was reported.
Time Frame: Up to Day 56
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV) | Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV
Number analyzed (Participants) | 160 | 172 | 188 | 360
Days | 4.5 [4.0 to 6.0] | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (2400mg IV); Test type: Superiority; p = 0.0218, Stratified Log Rank Test
Statistical Analysis 2: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): R10933+R10987 (8000mg IV); Test type: Superiority; p = 0.0156, Stratified Log Rank Test
Statistical Analysis 3: Comparison: Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Placebo vs Pooled (Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0067, Stratified Log Rank Test

31. Secondary Outcome: Pooled Analysis (Phases 1/2/3 [Cohort 1] and Phase 2 [Cohorts 1A/2/3]): Number of Participants With Treatment-Emergent Serious Adverse Events
Time Frame: Up to Day 169
Population: all FAS participants. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo: Participants received single dose of placebo matching to R10933+R10987 intravenously on Day 1
- Pooled R10933+R10987 2400 mg IV: Participants received a single dose of R10933+R10987 2400 mg intravenously on Day 1
- Pooled R10933+R10987 8000 mg IV: Participants received a single dose of R10933+R10987 8000 mg intravenously on Day 1.
- Pooled Combined R10933+R10987 IV: Participants received single dose of R10933+R10987 (2400 mg and 8000 mg) intravenously on Day 1
Arm/Group | Pooled Placebo | Pooled R10933+R10987 2400 mg IV | Pooled R10933+R10987 8000 mg IV | Pooled Combined R10933+R10987 IV
Number analyzed (Participants) | 730 | 740 | 733 | 1473
Participants | 203 | 177 | 181 | 358

32. Secondary Outcome: Pooled Analysis (Phases 1/2/3 [Cohort 1] and Phase 2 [Cohorts 1A/2/3]): Number of Participants With Grade >=2 Infusion Related Reactions up to Day 4
Time Frame: Up to Day 4
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Pooled R10933+R10987 2400 mg IV | Pooled R10933+R10987 8000 mg IV | Pooled Combined R10933+R10987 IV
Number analyzed (Participants) | 730 | 740 | 733 | 1473
Participants | 6 | 11 | 15 | 26

33. Secondary Outcome: Pooled Analysis (Phases 1/2/3 [Cohort 1] and Phase 2 [Cohorts 1A/2/3]): Number of Participants With Grade >=2 Hypersensitivity Reactions Up to Day 29
Time Frame: Up to Day 29
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Pooled R10933+R10987 2400 mg IV | Pooled R10933+R10987 8000 mg IV | Pooled Combined R10933+R10987 IV
Number analyzed (Participants) | 730 | 740 | 733 | 1473
Participants | 2 | 5 | 7 | 12

34. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Went on Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Description: Percentage of participants who went on mechanical ventilation in phase 3 (Cohort 1) and phase 2 (Cohort 1A) was reported.
Time Frame: by Day 29
Population: The seronegative mFAS was defined as all participants in mFAS with documented seronegative status at the baseline. As prespecified in protocol, separate analysis for placebo and R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3: Cohort 1 (Placebo): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Cohort 1
- Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Cohort 1.
- Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV): Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Cohort 1.
- Phase 3 (Cohort 1): Combined R10933+R10987 IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg or 8000mg intravenously on Day 1 in Cohort 1.
- Phase 2: Cohort 1A (Placebo): Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Cohort 1A.
- Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV): Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Cohort 1A.
- Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV): Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Cohort 1A
- Phase 2 (Cohort 1A): Combined R10933+R10987 IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg or 8000mg intravenously on Day 1 in Cohort 1A.
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 92 | 106 | 198
Percentage of Participants | 17.1 [9.2 to 28.0] | 8.8 [3.6 to 17.2] | 17.1 [9.7 to 27.0] | 13.0 [8.2 to 19.1] | 4.4 [1.2 to 11.0] | 3.3 [0.7 to 9.2] | 0.0 [0.0 to 0.0] | 1.5 [0.3 to 4.4]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.2162, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.8783, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.5583, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.7189, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0429, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.2103, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

35. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 6 Through Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died from Day 6 through Day 29 in phase 3 (cohort 1) and phase 2 (cohort 1A) were reported.
Time Frame: Day 6 to Day 29
Population: The seronegative mFAS was defined as all participants in mFAS with documented seronegative status at the baseline. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, separate analysis for placebo and R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3 (Cohort 1): Combined R10933+R10987 IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg or 8000 mg intravenously on Day 1 in Cohort 1.
- Phase 2 (Cohort 1A): Combined R10933+R10987 IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg or 8000 mg intravenously on Day 1 in Cohort 1A.
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 67 | 79 | 80 | 159 | 86 | 88 | 101 | 189
Percentage of Participants | 19.4 [10.8 to 30.9] | 6.3 [2.1 to 14.2] | 10.0 [4.4 to 13.6] | 8.2 [4.4 to 13.6] | 9.3 [4.1 to 17.5] | 3.4 [0.7 to 9.6] | 5.0 [1.6 to 11.2] | 4.2 [1.8 to 8.2]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0223, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.1256, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0230, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.1298, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.2642, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0970, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

36. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 1 Through Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died from Day 1 through Day 29 in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported.
Time Frame: Day 1 to Day 29
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 92 | 106 | 198
Percentage of Participants | 22.9 [13.7 to 34.4] | 7.5 [2.8 to 15.6] | 11.0 [5.1 to 19.8] | 9.3 [5.3 to 14.8] | 8.9 [3.9 to 16.8] | 3.3 [0.7 to 9.2] | 5.7 [2.1 to 11.9] | 4.5 [2.1 to 8.5]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0147, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0669, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0094, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.1306, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.3576, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.1476, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

37. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Were Discharged by Day 29 Based on Seronegative mFAS
Description: Percentage of participants who were discharged in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) by Day 29 were reported.
Time Frame: by Day 29
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 92 | 106 | 198
Percentage of Participants | 70.0 [57.9 to 80.4] | 85.0 [75.3 to 92.0] | 84.1 [74.4 to 91.3] | 84.6 [78.1 to 89.8] | 90.0 [81.9 to 95.3] | 94.6 [87.8 to 98.2] | 94.3 [88.1 to 97.9] | 94.4 [90.3 to 97.2]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0481, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0535, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0199, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.2784, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.2510, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.1702, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

38. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died or Were Readmitted to Hospital by Day 29 Based on Seronegative mFAS
Description: Percentage of participants who died or were readmitted to hospital in phase 3 (Cohort 1) and phase 2 (Cohort 1A) by Day 29 were reported. Readmission to hospital was based on investigator report.
Time Frame: Up to Day 29
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 92 | 106 | 198
Percentage of Participants | 27.1 [17.2 to 39.1] | 13.8 [7.1 to 23.3] | 14.6 [7.8 to 24.2] | 14.2 [9.2 to 20.5] | 22.2 [14.1 to 32.2] | 9.8 [4.6 to 17.8] | 11.3 [6.0 to 18.9] | 10.6 [6.7 to 15.8]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0500, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0663, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0229, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0208, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0388, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0092, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

39. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death up to Day 29 Based on Seronegative mFAS
Description: Percentage of participants with cumulative incidence of death in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) up to Day 29 from randomization were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: Up to Day 29
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Groups:
- Phase 2: Cohort 1A Combined R10933+R10987: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 (2400 mg or 8000 mg) intravenously on Day 1 in Cohort 1A.
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2: Cohort 1A Combined R10933+R10987
Number analyzed (Participants) | 51 | 70 | 70 | 140 | 70 | 78 | 90 | 168
Cumulative Incidence Percentage | 23.6 [15.1 to 35.6] | 7.8 [3.6 to 16.5] | 11.4 [6.1 to 20.7] | 9.6 [5.9 to 15.4] | 9.6 [4.9 to 18.3] | 3.6 [1.2 to 10.9] | 5.9 [2.7 to 12.8] | 4.8 [2.6 to 9.1]

40. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Description: Percentage of participants with cumulative incidence of mechanical ventilation in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) by Day 29 were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Groups:
- Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV): Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Cohort 1A
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 46 | 66 | 62 | 128 | 68 | 77 | 90 | 167
Cumulative Incidence Percentage | 18.2 [10.8 to 30.0] | 8.9 [4.4 to 17.8] | 17.6 [10.8 to 27.9] | 13.4 [8.9 to 19.8] | 4.7 [1.8 to 12.1] | 3.5 [1.1 to 10.5] | 0.0 [0.0 to 0.0] | 1.7 [0.5 to 5.1]

41. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death or Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Description: Percentage of participants with cumulative incidence of death or mechanical ventilation in Phase 3 (Cohort 1) and Phase 2 (Cohort 1A) by Day 29 were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: by Day 29
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 46 | 66 | 62 | 128 | 68 | 77 | 90 | 167
Cumulative Incidence Percentage | 30.4 [21.0 to 42.7] | 12.7 [7.0 to 22.3] | 21.2 [13.8 to 31.9] | 17.0 [12.0 to 23.8] | 11.8 [6.5 to 20.8] | 4.7 [1.8 to 12.1] | 5.9 [2.7 to 12.8] | 5.4 [2.9 to 9.7]

42. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Time to Discharge From Hospital Based on Seronegative mFAS
Description: Time to discharge from hospital up to Day 56 was reported.
Time Frame: Up to Day 56
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 86 | 99 | 198
Days | 8.5 [5.0 to 15.0] | 5.0 [4.0 to 7.0] | 6.0 [4.0 to 9.0] | 6.0 [4.0 to 7.0] | 4.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0370, stratified log-rank test
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.1596, stratified log-rank test
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0444, stratified log-rank test
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.1802, stratified log-rank test
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0407, stratified log-rank test
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0523, stratified log-rank test

43. Secondary Outcome: Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]: TWA Change From Baseline Viral Load (Seronegative mFAS) in NP Samples up to Day 11 Based on Seronegative mFAS
Description: TWA change from baseline in viral load up to Day 11 was calculated for each participant using the trapezoidal rule as the area under the curve for change from baseline at each time point divided by the time interval for the observation period. TWA change from baseline viral load in NP samples through Day 11, was measured by RT-qPCR in NP swab samples was reported. Baseline was defined as the last non-missing value measured prior to dosing. Negative changes indicate improvement in viral load.
Time Frame: Day 1 to Day 11
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 59 | 76 | 78 | 154 | 80 | 79 | 88 | 167
log10 copies/mL | -1.52 (0.17) | -2.03 (0.15) | -1.95 (0.15) | -2.00 (0.10) | -1.28 (0.14) | -1.88 (0.14) | -2.01 (0.14) | -1.95 (0.10)
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0245, ANCOVA
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0554, ANCOVA
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0179, ANCOVA
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0035, ANCOVA
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0003, ANCOVA
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0002, ANCOVA

44. Secondary Outcome: Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]: TWA Change From Baseline Viral Load (Seronegative mFAS) in NP Samples up to Day 29
Description: TWA change from baseline in viral load up to Day 29 was calculated for each participant using the trapezoidal rule as the area under the curve for change from baseline at each time point divided by the time interval for the observation period. TWA change from baseline viral load in NP samples through Day 29, was measured by quantitative RT-qPCR in NP swab samples was reported. Baseline was defined as the last non-missing value measured prior to dosing. Negative changes indicate improvement in viral load.
Time Frame: Day 1 to Day 29
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Groups:
- Phase 2 (Cohort 1A): Combined R10933+R10987 IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Cohort 1A.
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 64 | 77 | 79 | 156 | 84 | 82 | 93 | 175
log10 copies/mL | -2.72 (0.22) | -3.68 (0.20) | -3.69 (0.20) | -3.69 (0.14) | -2.66 (0.21) | -3.31 (0.21) | -3.58 (0.20) | -3.45 (0.14)
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0013, ANCOVA
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0010, ANCOVA
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0002, ANCOVA
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0250, ANCOVA
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0012, ANCOVA
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0014, ANCOVA

45. Secondary Outcome: Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]: Change From Baseline in Viral Load (Seronegative mFAS) as Measured by RT-qPCR in NP Swabs Over Time
Description: Change from baseline in viral load as measured by RT-qPCR in NP swabs over time was reported. Baseline was defined as the last non-missing value measured prior to dosing. Negative changes indicates improvement in viral load.
Time Frame: Days 3, 5, 7, 9, 11, 13, 15, 22 and 29
Population: The seronegative mFAS was defined as all participants in mFAS with documented seronegative status at the baseline. "Number of Participants Analyzed" = participants with measurements at baseline. "Number Analyzed" = participants with measurements for both baseline and the specific study day. As prespecified in protocol, separate analysis for placebo and R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 92 | 106 | 198
log10 copies/mL
  Change at Day 3: number analyzed (Participants) | 51 | 68 | 69 | 137 | 62 | 68 | 76 | 144
  Change at Day 3 | -1.10 (0.22) | -0.90 (0.19) | -0.93 (0.19) | -0.92 (0.14) | -0.85 (0.21) | -1.03 (0.20) | -1.41 (0.19) | -1.23 (0.14)
  Change at Day 5: number analyzed (Participants) | 46 | 62 | 54 | 116 | 50 | 44 | 53 | 97
  Change at Day 5 | -1.97 (0.27) | -2.28 (0.23) | -1.91 (0.25) | -2.11 (0.17) | -1.55 (0.25) | -2.21 (0.26) | -2.24 (0.24) | -2.21 (0.18)
  Change at Day 7: number analyzed (Participants) | 35 | 50 | 55 | 105 | 42 | 46 | 45 | 91
  Change at Day 7 | -1.97 (0.30) | -2.92 (0.26) | -3.22 (0.25) | -3.09 (0.18) | -2.29 (0.26) | -3.06 (0.25) | -3.49 (0.24) | -3.27 (0.17)
  Change at Day 9: number analyzed (Participants) | 33 | 52 | 49 | 101 | 36 | 42 | 49 | 91
  Change at Day 9 | -2.56 (0.32) | -3.89 (0.27) | -4.16 (0.27) | -4.03 (0.19) | -2.90 (0.28) | -3.75 (0.26) | -3.85 (0.24) | -3.80 (0.18)
  Change at Day 11: number analyzed (Participants) | 31 | 47 | 45 | 92 | 31 | 38 | 47 | 85
  Change at Day 11 | -3.22 (0.35) | -4.23 (0.29) | -4.57 (0.30) | -4.41 (0.21) | -3.88 (0.32) | -4.76 (0.30) | -4.34 (0.27) | -4.52 (0.2)
  Change at Day 13: number analyzed (Participants) | 29 | 45 | 47 | 92 | 37 | 43 | 50 | 93
  Change at Day 13 | -3.76 (0.35) | -5.18 (0.30) | -5.00 (0.29) | -5.10 (0.21) | -4.22 (0.31) | -4.56 (0.29) | -5.05 (0.27) | -4.82 (0.20)
  Change at Day 15: number analyzed (Participants) | 34 | 47 | 51 | 98 | 45 | 47 | 57 | 104
  Change at Day 15 | -4.42 (0.32) | -5.41 (0.28) | -5.25 (0.27) | -5.34 (0.19) | -4.14 (0.28) | -5.03 (0.27) | -5.23 (0.25) | -5.14 (0.18)
  Change at Day 22: number analyzed (Participants) | 28 | 47 | 47 | 94 | 36 | 40 | 53 | 93
  Change at Day 22 | -5.29 (0.30) | -5.74 (0.24) | -5.95 (0.24) | -5.85 (0.17) | -5.37 (0.30) | -5.75 (0.29) | -5.77 (0.25) | -5.75 (0.19)
  Change at Day 29: number analyzed (Participants) | 29 | 52 | 56 | 108 | 43 | 47 | 62 | 109
  Change at Day 29 | -5.90 (0.24) | -6.46 (0.18) | -6.60 (0.18) | -6.54 (0.13) | -5.77 (0.27) | -6.34 (0.26) | -6.36 (0.23) | -6.35 (0.17)
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Difference vs. Placebo by Day 29; Test type: Superiority; p = 0.0623, MMRM
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Difference vs. Placebo by Day 29; Test type: Superiority; p = 0.0203, MMRM
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Difference vs. Placebo by Day 29; Test type: Superiority; p = 0.0193, MMRM
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Difference vs. Placebo by Day 29; Test type: Superiority; p = 0.1206, MMRM
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Difference vs. Placebo by Day 29; Test type: Superiority; p = 0.0911, MMRM
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Difference vs. Placebo by Day 29; Test type: Superiority; p = 0.0645, MMRM

46. Secondary Outcome: Phase 3 [Cohort 1] and Phase 2 [Cohort 1A]: Percent Change From Baseline in Viral Load (Seronegative mFAS) as Measured by RT-qPCR in NP Swabs Over Time
Description: Percent change from baseline in viral load as measured by RT-qPCR in NP swabs over time was reported. Baseline was defined as the last non-missing value measured prior to dosing. Negative changes indicates improvement in viral load.
Time Frame: Days 3, 5, 7, 9, 11, 13, 15, 22 and 29
Population: The seronegative mFAS was defined as all participants in mFAS with documented seronegative status at the baseline. Number of Participants Analyzed" = participants with measurements at baseline. "Number Analyzed" = participants with measurements for both baseline and the specific study day. As prespecified in protocol, separate analysis for placebo and R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 70 | 80 | 82 | 162 | 90 | 92 | 106 | 198
Percent Change
  Percent change at Day 3: number analyzed (Participants) | 51 | 68 | 69 | 137 | 62 | 68 | 76 | 144
  Percent change at Day 3 | -92.04 [-97.12 to -78.01] | -87.52 [-94.82 to -69.93] | -88.15 [-95.07 to -71.52] | -87.94 [-93.51 to -77.61] | -85.92 [-94.47 to -64.12] | -90.65 [-96.19 to -77.01] | -96.15 [-98.37 to -90.90] | -94.15 [-96.86 to -89.09]
  Percent change at Day 5: number analyzed (Participants) | 46 | 62 | 54 | 116 | 50 | 44 | 53 | 97
  Percent change at Day 5 | -98.92 [-99.68 to -96.35] | -99.48 [-99.82 to -98.50] | -98.76 [-99.59 to -96.20] | -99.23 [-99.64 to -98.34] | -97.18 [-99.09 to -91.23] | -99.38 [-99.81 to -97.96] | -99.42 [-99.81 to -98.26] | -99.39 [-99.73 to -98.63]
  Percent change at Day 7: number analyzed (Participants) | 35 | 50 | 55 | 105 | 42 | 46 | 45 | 91
  Percent change at Day 7 | -98.92 [-99.73 to -95.76] | -99.88 [-99.96 to -99.62] | -99.94 [-99.98 to -99.82] | -99.92 [-99.96 to -99.82] | -99.49 [-99.84 to -98.36] | -99.91 [-99.97 to -99.73] | -99.97 [-99.99 to -99.90] | -99.95 [-99.98 to -99.88]
  Percent change at Day 9: number analyzed (Participants) | 33 | 52 | 49 | 101 | 36 | 42 | 49 | 91
  Percent change at Day 9 | -99.72 [-99.94 to -98.80] | -99.99 [-100.00 to -99.96] | -99.99 [-100.00 to -99.98] | -99.99 [-100.00 to -99.98] | -99.87 [-99.96 to -99.56] | -99.98 [-99.99 to -99.94] | -99.99 [-100.00 to -99.96] | -99.98 [-99.99 to -99.97]
  Percent change at Day 11: number analyzed (Participants) | 31 | 47 | 45 | 92 | 31 | 38 | 47 | 85
  Percent change at Day 11 | -99.94 [-99.99 to -99.70] | -99.99 [-100.00 to -99.98] | -100.00 [-100.00 to -99.99] | -100.00 [-100.00 to -99.99] | -99.99 [-100.00 to -99.94] | -100.00 [-100.00 to -99.99] | -100.00 [-100.00 to -99.98] | -100.00 [-100.00 to -99.99]
  Percent change at Day 13: number analyzed (Participants) | 29 | 45 | 47 | 92 | 37 | 43 | 50 | 93
  Percent change at Day 13 | -99.98 [-100.00 to -99.91] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -99.99 [-100.00 to -99.98] | -100.00 [-100.00 to -99.99] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Percent change at Day 15: number analyzed (Participants) | 34 | 47 | 51 | 98 | 45 | 47 | 57 | 104
  Percent change at Day 15 | -100.00 [-100.00 to -99.98] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -99.99 [-100.00 to -99.97] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Percent change at Day 22: number analyzed (Participants) | 28 | 47 | 47 | 94 | 36 | 40 | 53 | 93
  Percent change at Day 22 | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Percent change at Day 29: number analyzed (Participants) | 29 | 52 | 56 | 108 | 43 | 47 | 62 | 109
  Percent change at Day 29 | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Percent Difference vs. Placebo at Day 29; Test type: Superiority; p = 0.0623, MMRM
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Percent Difference vs. Placebo at Day 29; Test type: Superiority; p = 0.0203, MMRM
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Percent Difference vs. Placebo at Day 29; Test type: Superiority; p = 0.0193, MMRM
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Percent Difference vs. Placebo at Day 29; Test type: Superiority; p = 0.1206, MMRM
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Percent Difference vs. Placebo at Day 29; Test type: Superiority; p = 0.0911, MMRM
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Percent Difference vs. Placebo at Day 29; Test type: Superiority; p = 0.0645, MMRM

47. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Went on Mechanical Ventilation by Day 29 Based on High Viral Load mFAS
Description: as for outcome 34
Time Frame: by Day 29
Population: The High Viral Load mFAS was defined as all participants in mFAS with baseline SARS-CoV-2 viral load greater than (>) 10^6 copies per milliliter (mL). Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, separate analysis for placebo and R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 3 [Cohort 1] and Phase 2 [Cohort 1A].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 126 | 129 | 118 | 247 | 103 | 102 | 118 | 220
Percentage of Participants | 17.5 [11.3 to 25.2] | 8.5 [4.3 to 14.7] | 16.9 [10.7 to 25.0] | 12.6 [8.7 to 17.3] | 3.9 [1.1 to 9.6] | 2.9 [0.6 to 8.4] | 0.0 [0.0 to 0.0] | 1.4 [0.3 to 3.9]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0481, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.9880, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.2498, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.0457, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.2153, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

48. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 6 to Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who died in phase 3 (Cohort 1) and phase 2 (Cohort 1A) was reported.
Time Frame: Day 6 to Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 122 | 128 | 115 | 243 | 100 | 98 | 113 | 211
Percentage of Participants | 18.0 [11.7 to 26.0] | 10.2 [5.5 to 16.7] | 15.7 [9.5 to 23.6] | 12.8 [8.8 to 17.6] | 7.0 [2.9 to 13.9] | 3.1 [0.6 to 8.7] | 4.4 [1.5 to 10.0] | 3.8 [1.7 to 7.3]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0811, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.6701, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.2006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.3313, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.5542, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.2214, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

49. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died From Day 1 to Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who died in phase 3 (Cohort 1) and phase 2 (Cohort 1A) was reported.
Time Frame: Day 1 to Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 126 | 129 | 118 | 247 | 103 | 102 | 118 | 220
Percentage of Participants | 20.6 [13.9 to 28.8] | 10.9 [6.1 to 17.5] | 16.9 [10.7 to 25.0] | 13.8 [9.7 to 18.7] | 6.8 [2.8 to 13.5] | 2.9 [0.6 to 8.4] | 5.1 [1.9 to 10.7] | 4.1 [1.9 to 7.6]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0389, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.5208, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.1079, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.3315, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.5797, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.3036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

50. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Were Discharged by Day 29 Based on High Viral Load mFAS
Description: Percentage of participants who were discharged in phase 3 (Cohort 1) and phase 2 (Cohort 1A) was reported.
Time Frame: by Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 126 | 129 | 118 | 247 | 103 | 102 | 118 | 220
Percentage of Participants | 72.2 [63.5 to 79.8] | 83.7 [76.2 to 89.6] | 78.8 [70.3 to 85.8] | 81.4 [76.0 to 86.0] | 90.3 [82.9 to 95.2] | 96.1 [90.3 to 98.9] | 94.9 [89.3 to 98.1] | 95.5 [91.8 to 97.8]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0364, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.2795, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0588, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.0364, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.2795, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.0588, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

51. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Percentage of Participants Who Died or Were Readmitted to Hospital Over Time Based on High Viral Load mFAS
Description: Percentage of participants who died or were readmitted to hospital in phase 3 (Cohort 1) and phase 2 (Cohort 1A) over time were reported. Readmission to hospital was based on investigator report.
Time Frame: Up to Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 126 | 129 | 118 | 247 | 103 | 102 | 118 | 220
Percentage of Participants | 24.6 [17.4 to 33.1] | 18.6 [12.3 to 26.4] | 22.9 [15.7 to 31.5] | 20.6 [15.8 to 26.2] | 16.5 [9.9 to 25.1] | 10.8 [5.5 to 18.5] | 11.9 [6.6 to 19.1] | 11.4 [7.5 to 16.3]
Statistical Analysis 1: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.2635, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.8013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Phase 3: Cohort 1 (Placebo) vs Phase 3 (Cohort 1): Combined R10933+R10987 IV; Test type: Superiority; p = 0.4160, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV); Test type: Superiority; p = 0.2194, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV); Test type: Superiority; p = 0.3240, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Cohort 1A (Placebo) vs Phase 2 (Cohort 1A): Combined R10933+R10987 IV; Test type: Superiority; p = 0.1981, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

52. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death Over Time Based on High Viral Load mFAS
Description: Cumulative Incidence of Death Over Time in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: Up to Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 96 | 110 | 90 | 200 | 85 | 91 | 100 | 191
Cumulative Incidence Percentage | 21.1 [14.9 to 29.4] | 11.2 [6.8 to 18.2] | 17.9 [11.9 to 26.3] | 14.3 [10.5 to 19.5] | 7.2 [3.5 to 14.4] | 3.1 [1.0 to 9.4] | 5.3 [2.4 to 11.5] | 4.3 [2.3 to 8.2]

53. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Mechanical Ventilation Over Time Based on High Viral Load mFAS
Description: Cumulative Incidence of Mechanical Ventilation Over Time in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: Up to Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 87 | 104 | 83 | 187 | 83 | 90 | 100 | 190
Cumulative Incidence Percentage | 18.1 [12.3 to 26.2] | 8.8 [5.0 to 15.3] | 18.0 [12.0 to 26.5] | 13.1 [9.4 to 18.1] | 4.0 [1.5 to 10.4] | 3.1 [1.0 to 9.2] | 0.0 [0.0 to 0.0] | 1.5 [0.5 to 4.5]

54. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Cumulative Incidence of Death or Mechanical Ventilation Over Time Based on High Viral Load mFAS
Description: Cumulative Incidence of Death or Mechanical Ventilation Over Time in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported. Cumulative incidence percentage was estimated using Kaplan-Meier method.
Time Frame: Up to Day 29
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 87 | 104 | 83 | 187 | 83 | 90 | 100 | 190
Cumulative Incidence Percentage | 27.2 [20.2 to 35.9] | 15.0 [9.8 to 22.5] | 24.4 [17.6 to 33.4] | 19.5 [15.0 to 25.1] | 9.1 [4.9 to 16.8] | 4.1 [1.6 to 10.5] | 5.3 [2.4 to 11.5] | 4.8 [2.6 to 8.7]

55. Secondary Outcome: Phase 3 (Cohort 1) and Phase 2 (Cohort 1A): Time to Discharge Based on High Viral Load mFAS
Description: Time to Discharge in phase 3 (Cohort 1) and phase 2 (Cohort 1A) were reported.
Time Frame: Up to Day 56
Population: as for outcome 47
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3: Cohort 1 (Placebo) | Phase 3 (Cohort 1): R10933+R10987 (2400 mg IV) | Phase 3 (Cohort 1): R10933+R10987 (8000 mg IV) | Phase 3 (Cohort 1): Combined R10933+R10987 IV | Phase 2: Cohort 1A (Placebo) | Phase 2 (Cohort 1A): R10933+R10987 (2400 mg IV) | Phase 2 (Cohort 1A): R10933+R10987 (8000 mg IV) | Phase 2 (Cohort 1A): Combined R10933+R10987 IV
Number analyzed (Participants) | 126 | 129 | 118 | 247 | 103 | 102 | 118 | 220
days | 7.0 [5.0 to 10.0] | 7.0 [5.0 to 8.0] | 7.0 [5.0 to 8.0] | 7.0 [6.0 to 8.0] | 4.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.0] | 3.0 [3.0 to 3.0]

56. Secondary Outcome: Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Time-weighted Average (TWA) Change in Viral Load in Nasopharyngeal (NP) Samples Over Time Based on Seronegative mFAS
Description: Time-weighted average daily change over time up to Day 29 in viral load (log10 copies/mL), as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Up to Day 29
Population: Seronegative modified full analysis set (mFAS) = all participants in mFAS with documented seroneg status at baseline. "Number of Participants Analyzed" = participants with measurements at baseline. "Number Analyzed" = participants with measurements at both baseline and specific study day. As prespecified in protocol, pooled analysis of placebo and combined R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected/reported for Phase 1 [Cohort 1] and Phase 2 [Cohort 1].
Measure: Least Squares Mean (Standard Error); unit: log10 copies/milliliter (mL)
Groups:
- Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 Combined IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 (2400 mg and 8000 mg) intravenously on Day 1
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 Combined IV
Number analyzed (Participants) | 68 | 79 | 70 | 149
log10 copies/milliliter (mL)
  Time-weighted average change from baseline from Day 1 to Day 3: number analyzed (Participants) | 55 | 52 | 46 | 98
  Time-weighted average change from baseline from Day 1 to Day 3 | -0.33 (0.11) | -0.40 (0.11) | -0.60 (0.12) | -0.50 (0.08)
  Time-weighted average change from baseline from Day 1 to Day 5: number analyzed (Participants) | 58 | 57 | 52 | 109
  Time-weighted average change from baseline from Day 1 to Day 5 | -0.55 (0.14) | -0.86 (0.14) | -0.92 (0.14) | -0.89 (0.10)
  Time-weighted average change from baseline from Day 1 to Day 7: number analyzed (Participants) | 61 | 60 | 55 | 115
  Time-weighted average change from baseline from Day 1 to Day 7 | -0.70 (0.14) | -1.23 (0.14) | -1.23 (0.14) | -1.23 (0.10)
  Time-weighted average change from baseline from Day 1 to Day 9: number analyzed (Participants) | 61 | 61 | 57 | 118
  Time-weighted average change from baseline from Day 1 to Day 9 | -0.93 (0.16) | -1.47 (0.15) | -1.58 (0.16) | -1.52 (0.11)
  Time-weighted average change from baseline from Day 1 to Day 11: number analyzed (Participants) | 61 | 63 | 58 | 121
  Time-weighted average change from baseline from Day 1 to Day 11 | -1.12 (0.16) | -1.72 (0.16) | -1.78 (0.17) | -1.75 (0.12)
  Time-weighted average change from baseline from Day 1 to Day 13: number analyzed (Participants) | 61 | 64 | 58 | 122
  Time-weighted average change from baseline from Day 1 to Day 13 | -1.33 (0.18) | -1.96 (0.17) | -1.95 (0.18) | -1.96 (0.12)
  Time-weighted average change from baseline from Day 1 to Day 15: number analyzed (Participants) | 61 | 64 | 58 | 122
  Time-weighted average change from baseline from Day 1 to Day 15 | -1.50 (0.19) | -2.19 (0.18) | -2.16 (0.19) | -2.18 (0.13)
  Time-weighted average change from baseline from Day 1 to Day 22: number analyzed (Participants) | 61 | 64 | 58 | 122
  Time-weighted average change from baseline from Day 1 to Day 22 | -1.89 (0.22) | -2.62 (0.21) | -2.64 (0.22) | -2.63 (0.15)
  Time-weighted average change from baseline from Day 1 to Day 29: number analyzed (Participants) | 61 | 64 | 58 | 122
  Time-weighted average change from baseline from Day 1 to Day 29 | -2.35 (0.24) | -2.98 (0.23) | -2.95 (0.24) | -2.97 (0.17)

57. Secondary Outcome: Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Change From Baseline as Measured by RT-qPCR in NP Swabs Over Time Based on Seronegative mFAS
Description: as for outcome 45
Time Frame: Days 3, 5, 7, 9, 11, 13, 15, 22 and 29
Population: as for outcome 56
Measure: Least Squares Mean (Standard Error); unit: log10 copies/milliliter (mL)
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 Combined IV
Number analyzed (Participants) | 68 | 79 | 70 | 149
log10 copies/milliliter (mL)
  Time-weighted average change from baseline from Day 1 to Day 3: number analyzed (Participants) | 55 | 52 | 46 | 98
  Time-weighted average change from baseline from Day 1 to Day 3 | -0.66 (0.22) | -0.81 (0.21) | -1.08 (0.23) | -0.94 (0.16)
  Time-weighted average change from baseline from Day 1 to Day 5: number analyzed (Participants) | 47 | 43 | 40 | 83
  Time-weighted average change from baseline from Day 1 to Day 5 | -1.18 (0.26) | -2.08 (0.26) | -2.28 (0.27) | -2.18 (0.19)
  Time-weighted average change from baseline from Day 1 to Day 7: number analyzed (Participants) | 36 | 43 | 37 | 80
  Time-weighted average change from baseline from Day 1 to Day 7 | -1.62 (0.30) | -2.76 (0.27) | -2.56 (0.29) | -2.67 (0.20)
  Time-weighted average change from baseline from Day 1 to Day 9: number analyzed (Participants) | 27 | 32 | 31 | 63
  Time-weighted average change from baseline from Day 1 to Day 9 | -2.68 (0.34) | -3.24 (0.31) | -3.16 (0.32) | -3.20 (0.22)
  Time-weighted average change from baseline from Day 1 to Day 11: number analyzed (Participants) | 31 | 30 | 33 | 63
  Time-weighted average change from baseline from Day 1 to Day 11 | -3.55 (0.39) | -3.74 (0.38) | -3.94 (0.37) | -3.87 (0.26)
  Time-weighted average change from baseline from Day 1 to Day 13: number analyzed (Participants) | 25 | 31 | 23 | 54
  Time-weighted average change from baseline from Day 1 to Day 13 | -3.04 (0.38) | -5.01 (0.35) | -4.25 (0.39) | -4.68 (0.26)
  Time-weighted average change from baseline from Day 1 to Day 15: number analyzed (Participants) | 21 | 27 | 26 | 53
  Time-weighted average change from baseline from Day 1 to Day 15 | -4.60 (0.39) | -4.67 (0.35) | -5.01 (0.36) | -4.84 (0.25)
  Time-weighted average change from baseline from Day 1 to Day 22: number analyzed (Participants) | 18 | 28 | 26 | 54
  Time-weighted average change from baseline from Day 1 to Day 22 | -5.89 (0.37) | -5.21 (0.31) | -5.25 (0.32) | -5.23 (0.22)
  Time-weighted average change from baseline from Day 1 to Day 29: number analyzed (Participants) | 19 | 24 | 23 | 47
  Time-weighted average change from baseline from Day 1 to Day 29 | -6.01 (0.32) | -6.04 (0.27) | -6.16 (0.28) | -6.10 (0.20)

58. Secondary Outcome: Phase 1 [Cohort 1] and Phase 2 [Cohort 1]: Percentage of Participants Who Died or Went On Mechanical Ventilation by Day 29 Based on Seronegative mFAS
Time Frame: Through Day 29
Population: as for outcome 11
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of 2400mg or 8000 mg R10933+R10987 intravenously on Day 1
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 52 | 62 | 59 | 121
Percentage of Participants | 26.9 [19.0 to 34.8] | 17.7 [11.5 to 24.0] | 22.0 [15.1 to 28.9] | 19.8 [15.2 to 24.5]

59. Secondary Outcome: Phase 1 [Cohort 1] and Phase 2 [Cohort 1]: Percentage of Participants Who Died or Went On Mechanical Ventilation by Day 29 Based on High Viral Load mFAS
Time Frame: Through Day 29
Population: The High Viral Load mFAS was defined as all participants in mFAS with baseline SARS-CoV-2 viral load greater than (>) 10^6 copies per milliliter (mL). Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. As prespecified in protocol, separate analysis for placebo and R10933+R10987 IV (2400 mg and 8000 mg combined doses) were collected and reported for Phase 1 [Cohort 1] and Phase 2 [Cohort 1].
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Placebo | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (2400 mg IV) | Pooled (Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): R10933+R10987 (8000 mg IV) | Phase 1 [Cohort 1] and Phase 2 [Cohort 1]): Combined R10933+R10987 IV
Number analyzed (Participants) | 78 | 77 | 80 | 157
Percentage of Participants | 23.1 [17.0 to 29.2] | 23.4 [17.2 to 29.6] | 13.8 [8.8 to 18.7] | 18.5 [14.5 to 22.4]

60. Secondary Outcome: Phase 1 [Cohort 1]: Area Under the Concentration-Time Curve From Time 0 to 28 Days Post-dose (AUC0-28)
Time Frame: Up to Day 28
Population: Participants in Phase 1 (Cohort 1) who received any study drug of casirivimab and imdevimab and who had at least 1 non-missing drug concentration measurement following the first dose of study drug
Measure: Mean (Standard Deviation); unit: day*mg/L
Groups:
- Phase 1 [Cohort 1]: R10983+10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1
- Phase 1 [Cohort 1]: R10983+10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1
Arm/Group | Phase 1 [Cohort 1]: R10983+10987 2400mg IV | Phase 1 [Cohort 1]: R10983+10987 8000mg IV
Number analyzed (Participants) | 16 | 20
day*mg/L
  AUC0-28 of Casirivimab: number analyzed (Participants) | 9 | 12
  AUC0-28 of Casirivimab | 3026 (719) | 9678 (3362)
  AUC0-28 of Imdevimab: number analyzed (Participants) | 9 | 14
  AUC0-28 of Imdevimab | 2582 (581) | 8680 (2930)

61. Secondary Outcome: Concentration at the End of Infusion (Ceoi)
Time Frame: Day 1
Population: Participants who received any study drug of casirivimab and imdevimab
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Groups:
- Phase 1 [Cohort 1]: R10983+10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 1 [Cohort 1]: R10983+10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 2 (Cohort 1A): R10933+R10987 2400mg IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2 (Cohort 1A): R10933+R10987 8000mg IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2 (Cohort 1): R10933+R10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 1).
- Phase 2 (Cohort 1): R10933+R10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 1).
- Phase 2 (Cohort 2): R10933+R10987 2400mg IV: Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2 (Cohort 2): R10933+R10987 8000mg IV: Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2 (Cohort 3): R10933+R10987 2400mg IV: Participants on mechanical ventilation received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 2 (Cohort 3): R10933+R10987 8000mg IV: Participants on mechanical ventilation received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 3 (Cohort 1): R10933+R10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 3 (Cohort 1).
- Phase 3 (Cohort 1): R10933+R10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 3 (Cohort 1).
Arm/Group | Phase 1 [Cohort 1]: R10983+10987 2400mg IV | Phase 1 [Cohort 1]: R10983+10987 8000mg IV | Phase 2 (Cohort 1A): R10933+R10987 2400mg IV | Phase 2 (Cohort 1A): R10933+R10987 8000mg IV | Phase 2 (Cohort 1): R10933+R10987 2400mg IV | Phase 2 (Cohort 1): R10933+R10987 8000mg IV | Phase 2 (Cohort 2): R10933+R10987 2400mg IV | Phase 2 (Cohort 2): R10933+R10987 8000mg IV | Phase 2 (Cohort 3): R10933+R10987 2400mg IV | Phase 2 (Cohort 3): R10933+R10987 8000mg IV | Phase 3 (Cohort 1): R10933+R10987 2400mg IV | Phase 3 (Cohort 1): R10933+R10987 8000mg IV
Number analyzed (Participants) | 16 | 20 | 167 | 155 | 181 | 178 | 55 | 50 | 10 | 11 | 214 | 207
milligrams per liter (mg/L)
  Ceoi of Casirivimab: number analyzed (Participants) | 15 | 20 | 167 | 155 | 181 | 178 | 55 | 50 | 10 | 11 | 214 | 207
  Ceoi of Casirivimab | 231 (110) | 776 (372) | 272 (124) | 847 (300) | 288 (86.8) | 848 (261) | 286 (93.5) | 921 (262) | 284 (69.3) | 708 (128) | 307 (153) | 908 (338)
  Ceoi of Imdevimab: number analyzed (Participants) | 15 | 20 | 167 | 155 | 181 | 178 | 55 | 50 | 10 | 11 | 214 | 207
  Ceoi of Imdevimab | 243 (117) | 795 (371) | 283 (127) | 868 (298) | 300 (87.3) | 880 (268) | 302 (94.0) | 946 (244) | 290 (81.7) | 738 (124) | 312 (157) | 945 (351)

62. Secondary Outcome: Concentration at Day 28 (C28)
Time Frame: Day 28
Population: Participants who received any study drug of casirivimab and imdevimab and who had at least 1 non-missing drug concentration measurement following the first dose of study drug
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Phase 1 [Cohort 1]: R10983+10987 2400mg IV | Phase 1 [Cohort 1]: R10983+10987 8000mg IV | Phase 2 (Cohort 1A): R10933+R10987 2400mg IV | Phase 2 (Cohort 1A): R10933+R10987 8000mg IV | Phase 2 (Cohort 1): R10933+R10987 2400mg IV | Phase 2 (Cohort 1): R10933+R10987 8000mg IV | Phase 2 (Cohort 2): R10933+R10987 2400mg IV | Phase 2 (Cohort 2): R10933+R10987 8000mg IV | Phase 2 (Cohort 3): R10933+R10987 2400mg IV | Phase 2 (Cohort 3): R10933+R10987 8000mg IV | Phase 3 (Cohort 1): R10933+R10987 2400mg IV | Phase 3 (Cohort 1): R10933+R10987 8000mg IV
Number analyzed (Participants) | 9 | 9 | 91 | 96 | 91 | 93 | 25 | 26 | 3 | 5 | 149 | 146
mg/L
  C28 of Casirivimab | 50.7 (19.5) | 166 (108) | 64.8 (35.9) | 174 (65.1) | 50.0 (20.4) | 144 (89.8) | 26.4 (18.5) | 79.4 (61.4) | 9.06 (2.64) | 67.8 (31.1) | 49.1 (40.4) | 140 (66.1)
  C28 of Imdevimab | 36.1 (16.1) | 131 (84.1) | 54.7 (37.6) | 150 (62.9) | 39.8 (18.9) | 113 (68.8) | 18.7 (14.7) | 60.0 (53.9) | 5.25 (4.12) | 52.4 (24.7) | 40.8 (48.3) | 114 (62.6)

63. Secondary Outcome: Immunogenicity as Measured by Anti-drug Antibodies (ADAs) to REGN10933
Time Frame: Through Day 169
Population: ADA analysis set includes all treated participants from all phases/cohorts who received any amount of study drug and had at least one non-missing antibody variables result following the first dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled R10933+R10987 2400mg IV: Participants received a single 2400mg intravenous dose of R10933+R10987
- Pooled REGN10933+REGN10987 8000mg IV: Participants received a single 8000 mg intravenous dose of R10933+R10987
Arm/Group | Pooled Placebo | Pooled R10933+R10987 2400mg IV | Pooled REGN10933+REGN10987 8000mg IV
Number analyzed (Participants) | 503 | 504 | 497
Participants | 489 | 471 | 484

64. Secondary Outcome: Immunogenicity as Measured by Anti-drug Antibodies (ADAs) to REGN10987
Time Frame: Through Day 169
Population: as for outcome 63
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo: Participants received a single intravenous dose of placebo matching R10933+R10987
- Pooled R10933+R10987 2400mg IV: Participants received a single 2400mg dose of R10933+R10987 intravenously on Day 1
- Pooled REGN10933+REGN10987 8000mg IV: Participants received a single 8000 mg dose of R10933+R10987 intravenously on Day 1
Arm/Group | Pooled Placebo | Pooled R10933+R10987 2400mg IV | Pooled REGN10933+REGN10987 8000mg IV
Number analyzed (Participants) | 503 | 504 | 497
Participants | 467 | 444 | 463

65. Secondary Outcome: Immunogenicity as Measured by Neutralizing Antibody Status (NAb) to REGN10933
Time Frame: Through Day 57
Population: NAb analysis set includes all Phase 2/3 treated participants who received any study drug, had at least one non-missing antibody result following the first dose of study drug, and either tested negative at all ADA sampling times or tested positive for ADA with at least one non-missing NAb result after first dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled (Phase 2/3) Placebo: Participants received single dose of placebo matching to R10933+R10987 intravenously on Day 1
- Pooled (Phase 2/3) R10933+R10987 2400mg IV: Participants received a single 2400mg intravenous dose of R10933+R10987
- Pooled (Phase 2/3) REGN10933+REGN10987 8000mg IV: Participants received a single 8000 mg intravenous dose of R10933+R10987
Arm/Group | Pooled (Phase 2/3) Placebo | Pooled (Phase 2/3) R10933+R10987 2400mg IV | Pooled (Phase 2/3) REGN10933+REGN10987 8000mg IV
Number analyzed (Participants) | 503 | 504 | 497
Participants
  Anti-drug Antibody (ADA) Negative | 489 | 471 | 484
  Neutralizing antibody (NAb) Positive | 1 | 1 | 1

66. Secondary Outcome: Immunogenicity as Measured by Neutralizing Antibody Status (NAb) to REGN10987
Time Frame: Through Day 57
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled (Phase 2/3) Placebo | Pooled (Phase 2/3) R10933+R10987 2400mg IV | Pooled (Phase 2/3) REGN10933+REGN10987 8000mg IV
Number analyzed (Participants) | 503 | 504 | 497
Participants
  Anti-drug Antibody (ADA) Negative | 467 | 444 | 463
  Neutralizing antibody (NAb) Positive | 9 | 10 | 4

ADVERSE EVENTS:
Time Frame: From first dose of study drug to Day 169
Groups:
- Phase 1 Cohort 1: Placebo IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 1 Cohort 1: R10933+R10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 milligrams (mg) intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 1 Cohort 1: R10933+R10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 1 (Cohort 1).
- Phase 2 Cohort 1A: Placebo IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2 Cohort 1A: R10933+R10987 2400mg IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2 Cohort 1A: R10933+R10987 8000mg IV: Participants with COVID-19 symptoms but not requiring supplemental oxygen received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 1A).
- Phase 2 Cohort 1: Placebo IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 1).
- Phase 2 Cohort 1: R10933+R10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 1).
- Phase 2 Cohort 1: R10933+R10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 1).
- Phase 2 Cohort 2: Placebo IV: Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2 Cohort 2: R10933+R10987 2400mg IV: Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2 Cohort 2: R10933+R10987 8000mg IV: Participants on high-flow oxygen therapy but not on mechanical ventilation received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 2).
- Phase 2 Cohort 3: Placebo IV: Participants on mechanical ventilation received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 2 Cohort 3: R10933+R10987 2400mg IV: Participants on mechanical ventilation received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 2 Cohort 3: R10933+R10987 8000mg IV: Participants on mechanical ventilation received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 2 (Cohort 3).
- Phase 3 Cohort 1: Placebo IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of placebo matching to R10933+R10987 intravenously on Day 1 in Phase 3 (Cohort 1).
- Phase 3 Cohort 1: R10933+R10987 2400mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 2400 mg intravenously on Day 1 in Phase 3 (Cohort 1).
- Phase 3 Cohort 1: R10933+R10987 8000mg IV: Participants with O2 saturation > 93% on low-flow oxygen via nasal cannula, simple face mask, or other similar device received single dose of R10933+R10987 8000 mg intravenously on Day 1 in Phase 3 (Cohort 1).
Arm/Group | Phase 1 Cohort 1: Placebo IV | Phase 1 Cohort 1: R10933+R10987 2400mg IV | Phase 1 Cohort 1: R10933+R10987 8000mg IV | Phase 2 Cohort 1A: Placebo IV | Phase 2 Cohort 1A: R10933+R10987 2400mg IV | Phase 2 Cohort 1A: R10933+R10987 8000mg IV | Phase 2 Cohort 1: Placebo IV | Phase 2 Cohort 1: R10933+R10987 2400mg IV | Phase 2 Cohort 1: R10933+R10987 8000mg IV | Phase 2 Cohort 2: Placebo IV | Phase 2 Cohort 2: R10933+R10987 2400mg IV | Phase 2 Cohort 2: R10933+R10987 8000mg IV | Phase 2 Cohort 3: Placebo IV | Phase 2 Cohort 3: R10933+R10987 2400mg IV | Phase 2 Cohort 3: R10933+R10987 8000mg IV | Phase 3 Cohort 1: Placebo IV | Phase 3 Cohort 1: R10933+R10987 2400mg IV | Phase 3 Cohort 1: R10933+R10987 8000mg IV
All-Cause Mortality (participants affected / at risk) | 2/18 | 0/18 | 1/20 | 15/198 | 8/202 | 7/197 | 28/204 | 25/206 | 21/205 | 13/51 | 25/56 | 19/54 | 7/12 | 8/12 | 4/11 | 42/247 | 24/246 | 37/246
Serious Adverse Events (participants affected / at risk) | 3/18 | 3/18 | 2/20 | 43/198 | 29/202 | 32/197 | 63/204 | 47/206 | 47/205 | 20/51 | 31/56 | 26/54 | 9/12 | 11/12 | 5/11 | 65/247 | 56/246 | 69/246
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 1/20 | 0/198 | 0/202 | 0/197 | 0/204 | 0/206 | 0/205 | 0/51 | 0/56 | 0/54 | 0/12 | 1/12 | 1/11 | 0/247 | 1/246 | 2/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1: Placebo IV (N=18) | Phase 1 Cohort 1: R10933+R10987 2400mg IV (N=18) | Phase 1 Cohort 1: R10933+R10987 8000mg IV (N=20) | Phase 2 Cohort 1A: Placebo IV (N=198) | Phase 2 Cohort 1A: R10933+R10987 2400mg IV (N=202) | Phase 2 Cohort 1A: R10933+R10987 8000mg IV (N=197) | Phase 2 Cohort 1: Placebo IV (N=204) | Phase 2 Cohort 1: R10933+R10987 2400mg IV (N=206) | Phase 2 Cohort 1: R10933+R10987 8000mg IV (N=205) | Phase 2 Cohort 2: Placebo IV (N=51) | Phase 2 Cohort 2: R10933+R10987 2400mg IV (N=56) | Phase 2 Cohort 2: R10933+R10987 8000mg IV (N=54) | Phase 2 Cohort 3: Placebo IV (N=12) | Phase 2 Cohort 3: R10933+R10987 2400mg IV (N=12) | Phase 2 Cohort 3: R10933+R10987 8000mg IV (N=11) | Phase 3 Cohort 1: Placebo IV (N=247) | Phase 3 Cohort 1: R10933+R10987 2400mg IV (N=246) | Phase 3 Cohort 1: R10933+R10987 8000mg IV (N=246)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 7 (9) | 3 (3) | 7 (7) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 8 (8) | 5 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 2 (2) | 6 (6) | 10 (10) | 5 (5) | 0 (0) | 7 (7) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 11 (12) | 6 (6) | 5 (6)
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 9 (10) | 4 (4) | 6 (8) | 5 (6) | 4 (4) | 5 (6) | 1 (1) | 3 (3) | 0 (0) | 7 (8) | 7 (7) | 5 (5)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 7 (7) | 0 (0) | 6 (6) | 6 (6) | 4 (4) | 7 (7) | 4 (4) | 7 (7) | 8 (10) | 2 (2) | 1 (1) | 2 (2) | 10 (10) | 5 (5) | 8 (9)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burkholderia cepacia complex infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 7 (7)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Emphysematous cholecystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia serratia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 5 (6)
Serratia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral cardiomyopathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal tubular injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 2 (5) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 6 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECG signs of myocardial ischaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inflammatory marker increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mean arterial pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileostomy closure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1: Placebo IV (N=18) | Phase 1 Cohort 1: R10933+R10987 2400mg IV (N=18) | Phase 1 Cohort 1: R10933+R10987 8000mg IV (N=20) | Phase 2 Cohort 1A: Placebo IV (N=198) | Phase 2 Cohort 1A: R10933+R10987 2400mg IV (N=202) | Phase 2 Cohort 1A: R10933+R10987 8000mg IV (N=197) | Phase 2 Cohort 1: Placebo IV (N=204) | Phase 2 Cohort 1: R10933+R10987 2400mg IV (N=206) | Phase 2 Cohort 1: R10933+R10987 8000mg IV (N=205) | Phase 2 Cohort 2: Placebo IV (N=51) | Phase 2 Cohort 2: R10933+R10987 2400mg IV (N=56) | Phase 2 Cohort 2: R10933+R10987 8000mg IV (N=54) | Phase 2 Cohort 3: Placebo IV (N=12) | Phase 2 Cohort 3: R10933+R10987 2400mg IV (N=12) | Phase 2 Cohort 3: R10933+R10987 8000mg IV (N=11) | Phase 3 Cohort 1: Placebo IV (N=247) | Phase 3 Cohort 1: R10933+R10987 2400mg IV (N=246) | Phase 3 Cohort 1: R10933+R10987 8000mg IV (N=246)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT04426695/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT04426695/SAP_002.pdf